CLINICAL TRIAL: NCT00267371
Title: Effect of Septal Closure of Atrial PFO on Events of Migraine With Premere: ESCAPE Migraine Trial
Brief Title: ESCAPE Migraine Trial
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Insufficient enrollment
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1202-001; IDE G050112
Record Dates: First submitted 2005-12-16; First posted 2005-12-20 (Estimated); Last update posted 2019-02-04 (Actual); Status verified 2019-01

CONDITIONS: Migraine Disorders; Heart Septal Defects, Atrial
Keywords: Migraine headache; Patent Foramen Ovale; Patent Foramen Ovale Closure
MeSH Terms: conditions — Migraine Disorders; Heart Septal Defects, Atrial; Foramen Ovale, Patent

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Test Arm with Premere investigational (Active Comparator): PFO Closure with Premere investigational device.
  Interventions: Device: PFO Closure with Premere investigational device.
- Medical management/current medications (Active Comparator): Patients in the control group arm will not receive the medical device and will continue medical management.
  Interventions: Drug: Medical management/current medications per standard of care by personal physician.

INTERVENTIONS:
Device: PFO Closure with Premere investigational device. — PFO Closure with Premere investigational device.
  Arms: Test Arm with Premere investigational
Drug: Medical management/current medications per standard of care by personal physician. — Medical management with current medications per standard of care by personal physician.
  Other Names: Currently prescribed medications.
  Arms: Medical management/current medications

SUMMARY:
The purpose of this two arm controlled double-blind study is to determine the safety and effectiveness of PFO closure (closing a hole in the wall of the heart) in reducing the frequency of migraine headaches, in patients who experience migraine headaches and have a PFO, compared to medical therapy alone.

DETAILED DESCRIPTION:
Migraine headache is a neurological disorder characterized by chronic and disabling headache. Approximately 10-12% of humans, comprising some 28 million Americans, suffer from this disorder. Despite continual advances in medical management of migraine, many sufferers continue to experience frequent and disabling attacks despite appropriate medical therapy. Preventative medications, such as anti-epileptic drugs, anti-depressants, and beta-blockers, while effective for many patients, have side-effect profiles that preclude use in many patients. In the past decade, there has been growing evidence that patients with migraine, particularly those with aura, are more likely to have a patent foramen ovale.

A patent foramen ovale (PFO) is a persistent, flap-like opening in the wall of the heart, between the right and left atrium. Typically, this opening closes shortly after birth, however, in some people, it remains open.

While there is currently no proof for cause-effect relationship, several recent studies have confirmed a strong association between the presence of PFO and migraine with aura.

Comparison: This clinical study will compare PFO closure with medical therapy alone for the treatment of migraine headaches.

ELIGIBILITY:
Major Inclusion Criteria:

* Patient must be between the ages of 18 and 70;
* Patient must have a migraine history and demonstrate a refractoriness to medical treatment;
* Patient must have a Patent Foramen Ovale (PFO);
* Patient must be willing and able to give informed consent and complete required follow-up visits.

Major Exclusion Criteria:

* Patient has any medical condition or receives any medication that would preclude participation in the trial
* Patient is enrolled or intends to participate in another clinical study (of an investigational drug or device, new indication for an approved drug or device, or requirement of additional testing beyond standard clinical practice) during the study or within four weeks prior to his/her enrollment in the study.
* Patient is pregnant, or intends to become pregnant during the trial period

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2005-11; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Primary Endpoint 1: Effectiveness | 12 months
The primary effectiveness measure is the decrease in the frequency of migraine headaches. | monthly
The primary safety endpoint is the rate of major complications | monthly

SECONDARY OUTCOMES:
Secondary Endpoint 1: Effect of Aura | on-going
Secondary Endpoint 2: Assessment of Procedural Success and Long-Term Device Performance | Five years

CONTACTS AND LOCATIONS:
Overall Officials: Robert Sommer, MD, Principal Investigator — Columbia University; David Dodick, MD, Principal Investigator — Mayo Clinic
Locations (37):
- United States (37):
  - Mayo Clinic Hospital, Scottsdale, Arizona
  - Newport Beach Clinical Research Associates, Inc., Newport Beach, California
  - Sutter Institute for Medical Research, Sacramento, California
  - Alpine Clinical Research Center, Boulder, Colorado
  - Mile High Research Center, Denver, Colorado
  - Advanced Neurosciences Research, LLC, Fort Collins, Colorado
  - Hartford Headache Center, East Hartford, Connecticut
  - Medstar Clinical Research at Washington Hospital Center, Washington D.C., District of Columbia
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Neurology Associates, Maitland, Florida
  - Intercoastal Neurology, Sarasota, Florida
  - Axiom Clinical Research of Florida, Tampa, Florida
  - Neurology Specialists of Decatur, Decatur, Georgia
  - Evanston Northwestern HealthCare, Evanston, Illinois
  - Mid-Atlantic Headache Institute, Pikesville, Maryland
  - Stroke + NeuroCritical Care Stroke Service, Boston, Massachusetts
  - New England Regional Headache Center, Worcester, Massachusetts
  - Providence Hospital & Medical Centers, Inc., Southfield, Michigan
  - Mercy Health Research-Neurology, St Louis, Missouri
  - Radiant Research, St Louis, Missouri
  - Shore Neurology, PA, Toms River, New Jersey
  - Upstate Clinical Research, LLC, Albany, New York
  - MedARK Clinical Research, Morganton, North Carolina
  - Clinical Research of Winston-Salem, Winston-Salem, North Carolina
  - Wake Forest Univ. Health Sciences - BMC, Winston-Salem, North Carolina
  - Guilford Neurologic Associates, Inc., Winston-Salem, North Carolina
  - Neurology and Sleep Medicine, P.C., Bethlehem, Pennsylvania
  - Drexel University College of Medicine, Philadelphia, Pennsylvania
  - Clinical Trials Research Services, LLC, Pittsburgh, Pennsylvania
  - HAN Neurological Associates, Upland, Pennsylvania
  - Bellaire Neurology, PA, Bellaire, Texas
  - Texas Neurology, PA, Dallas, Texas
  - Houston Headache Clinic, Houston, Texas
  - University of Virginia Neurology, Charlottesville, Virginia
  - Commonwealth Clinical Research Specialists, Inc., Richmond, Virginia
  - Brighton Research Group, LLC, Virginia Beach, Virginia
  - Swedish Pain & Headache Specialist, Seattle, Washington

REFERENCES:
- [Derived] Sharan A, Huh B, Narouze S, Trentman T, Mogilner A, Vaisman J, Ordia J, Deer T, Venkatesan L, Slavin K. Analysis of adverse events in the management of chronic migraine by peripheral nerve stimulation. Neuromodulation. 2015 Jun;18(4):305-12; discussion 312. doi: 10.1111/ner.12243. Epub 2014 Oct 14. PMID 25313847